CLINICAL TRIAL: NCT03790631
Title: The OPTIMAL TDM Study: Determining Optimal Beta-lactam Plasma Concentrations Through Therapeutic Drug Monitoring
Acronym: OPTIMAL TDM
Status: Completed | Type: Observational
Sponsor: University of Geneva, Switzerland (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Angela HUTTNER, Principal Investigator, University of Geneva, Switzerland
Other Study IDs: 2018-01830
Record Dates: First submitted 2018-12-27; First posted 2018-12-31 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Beta-lactam Antibiotics; Therapeutic Drug Monitoring; Toxicity; Efficacy; Imipenem; Meropenem; Piperacillin; Flucloxacillin; Amoxicillin; Ceftazidime; Cefepime

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (7):
- imipenem TDM: Adult patients receiving imipenem for suspected or confirmed bacterial infection. TDM will be performed to assess intermediate and trough levels once the patient is at steady-state.
  Interventions: Other: The study is observational.
- meropenem TDM: Adult patients receiving meropenem for suspected or confirmed bacterial infection. TDM will be performed to assess intermediate and trough levels once the patient is at steady-state.
  Interventions: Other: The study is observational.
- piperacillin TDM: Adult patients receiving piperacillin (with or without tazobactam) for suspected or confirmed bacterial infection. TDM will be performed to assess intermediate and trough levels once the patient is at steady-state.
  Interventions: Other: The study is observational.
- flucloxacillin TDM: Adult patients receiving flucloxacillin for suspected or confirmed bacterial infection. TDM will be performed to assess intermediate and trough levels once the patient is at steady-state.
  Interventions: Other: The study is observational.
- amoxicillin TDM: Adult patients receiving amoxicillin for suspected or confirmed bacterial infection. TDM will be performed to assess intermediate and trough levels once the patient is at steady-state.
  Interventions: Other: The study is observational.
- ceftazidime TDM: Adult patients receiving ceftazidime for suspected or confirmed bacterial infection. TDM will be performed to assess intermediate and trough levels once the patient is at steady-state.
  Interventions: Other: The study is observational.
- cefepime TDM: Adult patients receiving cefepime for suspected or confirmed bacterial infection. TDM will be performed to assess intermediate and trough levels once the patient is at steady-state.
  Interventions: Other: The study is observational.

INTERVENTIONS:
Other: The study is observational. — The study is observational.

SUMMARY:
Little is known of beta-lactam antibiotics' true therapeutic plasma concentration range. The aims of this study are to define evidence-based, safe and effective upper and lower limits of the plasma concentrations of imipenem, meropenem, amoxicillin, flucloxacillin, piperacillin, ceftazidime and cefepime in patients at increased risk of serious bacterial infections and currently understudied pharmacokinetics (the critically ill, the elderly, and the immunosuppressed).

This prospective observational study will include adult patients with suspected or confirmed systemic bacterial infection receiving one of the above-named antibiotics and hospitalized in intensive-care, step-down, or hematology-oncology units of the Geneva University Hospitals (HUG).

Eligible patients will be identified via the electronic health record (EHR). Patients receiving traditional intermittent dosing or prolonged infusions will undergo TDM for at least one intermediate (mid-interval) and one trough level at 24 hours (-12 or +48 hours) after the therapy's start. Patients receiving continuous infusions will undergo TDM for at least one steady-state level. Clinical course will be observed for 30 days from the start of the study antibiotic (1st day of study antibiotic =day 1).

The primary outcome is incidence of clinical toxicity through day 30 after start of study antibiotic (as stratified by BL trough concentration). Secondary outcomes are listed below.

DETAILED DESCRIPTION:
Little is known of beta-lactam antibiotics' true therapeutic plasma concentration range. The aims of this study are to define evidence-based, safe and effective upper and lower limits of the plasma concentrations of imipenem, meropenem, amoxicillin, flucloxacillin, piperacillin, ceftazidime and cefepime in patients at increased risk of serious bacterial infections and currently understudied pharmacokinetics (the critically ill, the elderly, and the immunosuppressed).

This prospective observational study will include adult patients with suspected or confirmed systemic bacterial infection receiving one of the above-named antibiotics and hospitalized in intensive-care, step-down, or hematology-oncology units of the Geneva University Hospitals (HUG).

Eligible patients will be identified via the electronic health record (EHR). Patients receiving traditional intermittent dosing or prolonged infusions will undergo TDM for at least one intermediate (mid-interval) and one trough level at 24 hours (-12 or +48 hours) after the therapy's start. Patients receiving continuous infusions will undergo TDM for at least one steady-state level. Clinical course will be observed for 30 days from the start of the study antibiotic (1st day of study antibiotic =day 1).

The primary outcome is incidence of clinical toxicity through day 30 after start of study antibiotic (as stratified by BL trough concentration). Secondary outcomes are listed below.

ELIGIBILITY:
Inclusion Criteria:

- Hospitalized patients with suspected or confirmed systemic bacterial infection:

1. Receiving either imipenem-cilastatin, meropenem, amoxicillin (±clavulanic acid), flucloxacillin, piperacillin-tazobactam, ceftazidime or cefepime
2. Aged ≥18 years
3. Requiring intensive or intermediate-intensive (step-down) care OR severely immunosuppressed (see definitions)

Exclusion Criteria:

1. Planned imminent transfer to an outside hospital
2. Poor prognosis with life expectancy <1 week and/or intended transition to palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included patients will be adults (≤18 years) hospitalized in the intensive-care, step-down, or hematology-oncology units of the Geneva University Hospitals and treated with one of the above-listed 7 beta-lactam antibiotics for a suspected or confirmed bacterial infections.
Sampling Method: Non-Probability Sample
Enrollment: 771 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of clinical toxicity through day 30 after start of study antibiotic | day 30 after start of antibiotic
  Incidence of clinical toxicity through day 30 after start of study antibiotic (as stratified by BL trough concentration)

SECONDARY OUTCOMES:
Clinical response: incidence of clinical cure | day 30
  Clinical response to therapy through day 30 will be measured study-wide. "Clinical response" is either clinical cure (resolution of symptoms) or clinical failure (lack of improvement in signs and symptoms of infection OR recurrence of signs/symptoms of infection after initial improvement OR death in the 30-day study period considered at least possibly due to the infection). Where the MIC is unavailable, EUCAST epidemiologic cutoffs (ECOFF) will be used; if no organism is isolated, non-species-related breakpoints for targeted organisms (e.g., Pseudomonas aeruginosa) will be used.
clinical response in patients with neutropenic fever: incidence of clinical cure in this subpopulation | day 30
  Clinical response (as in outcome no. 2) in the subgroup of patients with neutropenic fever at the time of BL therapy. ("Clinical response" is either clinical cure (resolution of symptoms) or clinical failure (lack of improvement in signs and symptoms of infection OR recurrence of signs/symptoms of infection after initial improvement OR death in the 30-day study period considered at least possibly due to the infection).)
30-day mortality attributable to the treated infection | day 30
  30-day mortality attributable to the treated infection
30-day all-cause mortality | day 30
  30-day all-cause mortality
incidence of reversible toxicity | day 30
  Proportion of adverse events (AE) that are reversible after discontinuation of the relevant BL antibiotic
Incidence of Clostridium difficile infection | day 30
  Incidence of Clostridium difficile infection
Incidence of clinical toxicity of piperacillin-tazobactam when co-administered with vancomycin | day 30
  Incidence of clinical toxicity of piperacillin-tazobactam (and other beta-lactam antibiotics) when co-administered with vancomycin
Incidence of emergence of resistance | day 30
  Prevalence of emerging resistance to study antibiotics in clinical isolates (from baseline)
Incidence of undetectable beta-lactam plasma concentrations | day 30
  Proportion of patients with undetectable beta-lactam trough and/or intermediate concentrations
Incidence of off-label prescribing | day 30
  Proportion of patients for whom (a) beta-lactam dosing is "off-label" according to Swiss recommendations and (b) there are no dosing recommendations (e.g., hemofiltration)
The correlation of free versus total flucloxacillin concentrations | day 30
  The correlation of free versus total flucloxacillin concentrations (in a subset of patients, free flucloxacillin plasma levels will also be measured and compared to those of total flucloxacillin).
Median intermediate and trough plasma concentrations of tazobactam | through day 30
  In a subset of patients receiving piperacillin/tazobactam, median intermediate and trough plasma concentrations of tazobactam (beta-lactamase inhibitor) in proportion to piperacillin in patients receiving piperacillin-tazobactam
Beta-lactam trough concentration/minimal inhibitory concentration (MIC) index | day 1 (±1)
  The trough beta-lactam (BL) concentration/minimal inhibitory concentration (MIC) index on day 1 (±1) will be measured in all patients for later correlation analyses with clinical outcomes (clinical success versus failure).

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Data may be housed in a publicly accessible, non-profit digital repository such as Dryad or EUDAT.

REFERENCES:
- [Background] Bricheux A, Lenggenhager L, Hughes S, Karmime A, Lescuyer P, Huttner A. Therapeutic drug monitoring of imipenem and the incidence of toxicity and failure in hospitalized patients: a retrospective cohort study. Clin Microbiol Infect. 2019 Mar;25(3):383.e1-383.e4. doi: 10.1016/j.cmi.2018.11.020. Epub 2018 Dec 4. PMID 30528370
- [Background] Huwyler T, Lenggenhager L, Abbas M, Ing Lorenzini K, Hughes S, Huttner B, Karmime A, Uckay I, von Dach E, Lescuyer P, Harbarth S, Huttner A. Cefepime plasma concentrations and clinical toxicity: a retrospective cohort study. Clin Microbiol Infect. 2017 Jul;23(7):454-459. doi: 10.1016/j.cmi.2017.01.005. Epub 2017 Jan 19. PMID 28111294
- [Background] Muller AE, Huttner B, Huttner A. Therapeutic Drug Monitoring of Beta-Lactams and Other Antibiotics in the Intensive Care Unit: Which Agents, Which Patients and Which Infections? Drugs. 2018 Mar;78(4):439-451. doi: 10.1007/s40265-018-0880-z. PMID 29476349
- [Background] Huttner A, Harbarth S, Hope WW, Lipman J, Roberts JA. Therapeutic drug monitoring of the beta-lactam antibiotics: what is the evidence and which patients should we be using it for? J Antimicrob Chemother. 2015 Dec;70(12):3178-83. doi: 10.1093/jac/dkv201. Epub 2015 Jul 17. PMID 26188037
- [Derived] Marti C, Stirnemann J, Lescuyer P, Tonoli D, von Dach E; OPTIMAL TDM Study Group; Huttner A. Therapeutic drug monitoring and clinical outcomes in severely ill patients receiving amoxicillin: a single-centre prospective cohort study. Int J Antimicrob Agents. 2022 Jun;59(6):106601. doi: 10.1016/j.ijantimicag.2022.106601. Epub 2022 May 6. PMID 35533793